CLINICAL TRIAL: NCT00867607
Title: A Double-blind, Vehicle-controlled Study to Assess the Safety, Tolerability, and Efficacy of Three Weeks of Daily Dermal Application of MRX-6 (2% HyPE) on the Treatment of Mild to Moderate Contact Dermatitis of the Hand and Forearm
Brief Title: Safety, Tolerability, and Efficacy of 21 Days Dermal Application of MRX-6 on Mild to Moderate Contact Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Morria Biopharmaceuticals PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRX6-201ver4-HMO-CTIL
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2012-03

CONDITIONS: Allergic Contact Dermatitis
Keywords: Contact dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Allergic Contact; Dermatitis, Contact; Eczema | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MRX-6 (2%) (Experimental)
  Interventions: Drug: MRX-6
- MRX-6 (1%) (Experimental)
  Interventions: Drug: MRX-6
- MRX-6 (0.2%) (Experimental)
  Interventions: Drug: MRX-6
- Steroid (Active Comparator)
  Interventions: Drug: Steroid

INTERVENTIONS:
Drug: MRX-6 — b.i.d treatment for 21 days
  Arms: MRX-6 (0.2%); MRX-6 (1%); MRX-6 (2%)
Drug: Steroid — b.i.d. 21 days
  Arms: Steroid

SUMMARY:
A Double-blind, Vehicle-controlled Study to Assess the Safety, Tolerability, and Efficacy of Three Weeks of Daily Dermal Application of MRX-6 or steroid on the Treatment of Mild to Moderate Allergic Contact Dermatitis of the Hand and Forearm.

Total number of patients: up to 80.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women between 18 and 65 years old.
2. Male or non-pregnant female subjects who agree to comply with applicable contraceptive requirements of the protocol. Details on potential child-bearing status, methods to regularly exclude pregnancy throughout the study and acceptable forms of contraception are provided in Section 3.4.1 of the protocol.
3. Satisfactory medical assessment with no clinically significant and relevant abnormalities (of medical history, physical examination, clinical or laboratory evaluation [hematology, biochemistry, urinalysis]) as determined by the Principal Investigator, that might interfere with the assessment of the subjects dermatitis or the assessment of the safety or efficacy of the Study Drug.
4. The subject must understand and be able, willing and likely to fully comply with study procedures and restrictions.
5. Subject can understand and provide written informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related procedures listed in Section 5.1.1 of the protocol.
6. Subject has mild to moderate bilateral allergic contact dermatitis on each hand, possibly extending to the forearm, according to Physicians Visual Assessment as described in Section 5.2.1 of the protocol. Mild to moderate disease is considered a PVA score of 10 or greater and there should be no more than a 1-point difference between hands.
7. Have a + reaction to the Standard European Series patch testing kit (Chemotechnique Diagnostics Products, Malmo, Sweden) after application for 2 days, as described in Section 5.2.2 of the protocol.

Exclusion Criteria:

1. Current or recurrent disease that could affect the action, absorption or disposition of the Study Drug, or clinical or laboratory assessments.
2. Have used topical antihistamines in the past 2 weeks, topical corticosteroids or received Psoralen plus ultra violet light therapy (PUVA) in the past 4 weeks, or have taken oral retinoids, corticosteroids in the past 8 weeks (inhaled or intranasal corticosteroids are allowed, if stable dose).
3. Use of any prescription or OTC medication (excluding hormonal contraceptive, hormonal replacement therapy, inhaled or intranasal corticosteroids , or oral NSAIDs) that, in the opinion of the Principal Investigator, could affect (improve or worsen) the condition being studied, or could affect the action, absorption or disposition of the Study Drug, or clinical or laboratory assessments.
4. Patients must not have used another investigational product or taken part in a clinical trial within the last 30 days prior to enrolment.
5. Female patients who are pregnant or lactating, including females with a positive pregnancy test at screening, must be excluded.
6. The subject known to have a positive hepatitis virus test (Hepatitis B virus surface antigen or hepatitis C virus antibody) or a positive human immunodeficiency virus (HIV) antibody test.
7. A history of hypersensitivity to any of the Study Drugs or their excipients.
8. Subject has any other significant dermatological condition that affects >10% of the body surface area or general medical condition that could interfere with the study evaluation
9. Subject has any significant medical condition that could compromise immune responsiveness
10. Subject has a history of alcoholism or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of three dose levels of topical MRX-6 (0.2%, 1.0% and 2% HyPE) when administered twice daily (b.i.d.) for 21 consecutive days | Day 21

SECONDARY OUTCOMES:
Difference in percentage change in each subject's total Physician's Visual Assessment (PVA) score from Baseline to Day 21 between the vehicle and MRX-6 treated hands/forearms. | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Ramot, MD, Principal Investigator — Hadassah university hospital, Jerusalem Israel
Locations (2):
- Israel (2):
  - dermatology department, Hadassah university hospital, Jerusalem, Israel
  - Department of Dermatology, Hadassah Hospital, Ein Karem, Jerusalem

REFERENCES:
- [Result] Ingber A, Cohen Y, Krimsky M, Yedgar S. A novel treatment of contact dermatitis by topical application of phospholipase A2 inhibitor: a double-blind placebo-controlled pilot study. Int J Immunopathol Pharmacol. 2007 Jan-Mar;20(1):191-5. doi: 10.1177/039463200702000123. PMID 17346444